CLINICAL TRIAL: NCT05661994
Title: Effects of Omega-3 Fatty Acid Supplementation on Serum Fetuin-A Levels in Patients With Coronary Artery Disease
Brief Title: Omega-3 Supplementation on Serum Fetuin-A Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Mehmet Arif Icer, Principal Investigator, Amasya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 66175679-514.11.01-E.290378
Record Dates: First submitted 2022-10-31; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Coronary Artery Disease
Keywords: Fetuin-A; Omega-3 fatty acid; Coronary artery disease; Nutrient intake
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients with CAD were divided into the "Omega-3 Group (n:16)" and "Control Group (n:18)". Low-fat diet principles were explained to both groups at baseline. While 1.560 mg/day omega-3 FA supplementation was given to the patients in the omega-3 group for eight weeks, but not in the control group.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omega-3 Group (Experimental): While 1.560 mg/day omega-3 FA supplementation was given to the patients in the omega-3 group for eight weeks, but not in the control group.
  Interventions: Dietary Supplement: Omega-3 fatty acid supplementation
- Control Group (No Intervention): While 1.560 mg/day omega-3 FA supplementation was given to the patients in the omega-3 group for eight weeks, but not in the control group.

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acid supplementation — Patients with CAD were divided into the "Omega-3 Group (n:16)" and "Control Group (n:18)" to evaluate the effects of omega-3 FA supplementation on biochemical parameters, especially serum fetuin-A, anthropometric measurements, and nutritional status. 1.560 mg/day omega-3 FA supplementation was applied for 8 weeks to 16 participants with CAD included in the omega-3 group.
  Arms: Omega-3 Group

SUMMARY:
Background and aims: One of the investigated possible modulators of serum fetuin-A, associated with the risk of developing coronary artery disease (CAD), is omega-3 fatty acids (FAs). This study aims to evaluate the effects of omega-3 FA supplementation on serum fetuin-A concentration in patients with CAD.

Methods: The study was carried out on 34 male volunteer patients aged 35-75 years, newly diagnosed with CAD by conventional coronary angiography. Patients with CAD were divided into the "Omega-3 Group (n:16)" and "Control Group (n:18)". Low-fat diet principles were explained to both groups at baseline. While 1.560 mg/day omega-3 FA supplementation was given to the patients in the omega-3 group for eight weeks, but not in the control group. Food intake was recorded using six-day food records.

DETAILED DESCRIPTION:
The study was carried out on 34 male volunteer patients aged 35-75 years, newly diagnosed with coronary artery disease (CAD) by conventional coronary angiography. The study did not include the individuals who have dieted in the last six months, been taking an omega-3 FA and/or vitamin/mineral supplements or statin group drugs, been BMI <18.5 and ≥40 kg/m2, been fasting blood glucose ≥ 126 mg/dL, had a systemic disease such as Type 1 and Type 2 diabetes, kidney diseases, liver diseases, cancer and neurological diseases, active athletes, regular exercisers. Gazi University Faculty of Medicine Clinical Research Ethics Committee approved the study on 26 November 2020 with approval number 810. In addition, the necessary approval was obtained from the Turkish Medicines and Medical Devices Agency with the decision numbered 66175679-514.11.01-E.290378. All participants gave signed informed consent and the study was conducted in accordance with Helsinki Declaration.

Patients with CAD were divided into the "Omega-3 Group (n:16)" and "Control Group (n:18)" to evaluate the effects of omega-3 FA supplementation on biochemical parameters, especially serum fetuin-A, anthropometric measurements, and nutritional status. 1.560 mg/day omega-3 FA supplementation was applied for 8 weeks to 16 participants with CAD included in the omega-3 group, and the principles of a low-fat diet were explained. The principles of the low-fat diet without omega-3 FA supplementation were explained to 18 participants with CAD in the control group. The data of the participants were collected at the beginning, every 15 days and at the end of the 8th week.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteer patients aged 35-75 years
* Patients with newly diagnosed with coronary artery disease by conventional coronary angiography

Exclusion Criteria:

* Individuals who have dieted in the last six months
* Use of omega-3 fatty acid and/or vitamin/mineral supplements or statin group drugs
* BMI <18.5 and ≥40 kg/m2
* Fasting blood glucose ≥ 126 mg/dL
* Presence of systemic diseases such as Type 1 and Type 2 diabetes, kidney diseases, liver diseases, cancer or neurological diseases
* Active athletes and/or those who exercise regularly

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Analysis of serum total cholesterol (mg/dL), low-density lipoprotein cholesterol (LDL-C) (mg/dL), high-density lipoprotein cholesterol (HDL-C) (mg/dL), triglyceride (mg/dL), fasting blood glucose (mg/dL), calcium (mg/dL) and phosphorus (mg/dL) | 8 weeks
  The blood samples of the participants were taken by the nurse after 8 hours of fasting for the analysis of biochemical parameters. The blood samples of the participants were analyzed at the beginning and at the end of the 8th week in the biochemistry laboratory of the Faculty of Medicine, Gazi University to determine total cholesterol (mg/dL), low-density lipoprotein cholesterol (LDL-C) (mg/dL), high-density lipoprotein cholesterol (HDL-C) (mg/dL), triglyceride (mg/dL), fasting blood glucose (mg/dL), calcium (mg/dL) and phosphorus (mg/dL) levels of the participants.
Analysis of serum adiponectin (µg/mL) | 8 weeks
  The blood samples of the participants were taken by the nurse after 8 hours of fasting for the analysis of biochemical parameters. Adiponectin (µg/mL) concentrations in blood samples were analyzed in a private laboratory.
  For the analysis of adiponectin, blood samples taken into yellow-capped gel tubes were kept at room temperature for 30-45 minutes while the tubes were in an upright position, then centrifuged at 3,000 rpm for 15 min and the serum was frozen at -80°C until assayed.
Analysis of serum C-reactive protein (CRP) (mg/L) | 8 weeks
  The blood samples of the participants were taken by the nurse after 8 hours of fasting for the analysis of biochemical parameters. The blood samples of the participants were analyzed at the beginning and at the end of the 8th week in the biochemistry laboratory of the Faculty of Medicine, Gazi University to determine serum C-reactive protein (CRP) (mg/L) levels of the participants.
Analysis of serum fasting insulin (µIU/mL) | 8 weeks
  The blood samples of the participants were taken by the nurse after 8 hours of fasting for the analysis of biochemical parameters. The blood samples of the participants were analyzed at the beginning and at the end of the 8th week in the biochemistry laboratory of the Faculty of Medicine, Gazi University to determine serum fasting insulin (µIU/mL) levels of the participants.
Analysis of serum high-sensitivity troponin T (hs) -TnT) (ng/mL) | 8 weeks
  The blood samples of the participants were taken by the nurse after 8 hours of fasting for the analysis of biochemical parameters. The blood samples of the participants were analyzed at the beginning and at the end of the 8th week in the biochemistry laboratory of the Faculty of Medicine, Gazi University to determine serum high-sensitivity troponin T (hs) -TnT) (ng/mL) levels of the participants.
Analysis of serum fetuin-A (ng/mL) | 8 weeks
  The blood samples of the participants were taken by the nurse after 8 hours of fasting for the analysis of biochemical parameters. Fetuin-A (ng/mL) concentrations in blood samples were analyzed in a private laboratory.
  For the analysis of fetuin-A levels, blood samples taken into yellow-capped gel tubes were kept at room temperature for 30-45 minutes while the tubes were in an upright position, then centrifuged at 3,000 rpm for 15 min and the serum was frozen at -80°C until assayed.
Homeostatic model assessment-insulin resistance (HOMA-IR) | 8 weeks
  Homeostatic model assessment-insulin resistance (HOMA-IR) values were calculated according to the formula: fasting insulin (mIU/mL) × fasting glucose (mg/dL)/405.
Nutritional assessment | 8 weeks
  A total of six-day food records (three-day food records with a 24-hour dietary recall method every 15 days and three consecutive-day food records at week 8.) were taken by the researcher for determining participants' daily dietary energy and nutrient intake. The energy and nutrient intake was calculated using the Nutrition Information System (BeBiS) program.
Body weight analysis | 8 weeks
  The body weight of the participants was analyzed at the beginning, every 15 days and at the end of the 8th week. The body weight of the participants was analyzed through Tanita BC 601 bio-electric impedance device after 10-12 hours of hunger.
Height and waist circumferences (cm) measurement | 8 weeks
  The height and waist circumferences (cm) of the participants were measured by using a non-elastic tape measure.
Body mass index calculation | 8 weeks
  Body mass indexes were calculated by applying 'body weight/height2 (kg/m2)' equation.
Body fat percentage (%) and body water percentage (%) analysis | 8 weeks
  The body fat percentage and body water percentage of the participants were analyzed at the beginning, every 15 days and at the end of the 8th week. The body fat percentage and body water percentage of the participants were analyzed through Tanita BC 601 bio-electric impedance device after 10-12 hours of hunger.
Body muscle mass analysis | 8 weeks
  The body muscle mass of the participants was analyzed at the beginning, every 15 days and at the end of the 8th week. The body muscle mass of the participants was analyzed through Tanita BC 601 bio-electric impedance device after 10-12 hours of hunger.

SECONDARY OUTCOMES:
Personal Information Form | 8 weeks
  The data of the study were collected using a face-to-face interview technique through a questionnaire. Descriptive information about the individuals (age, gender, marital status, education level, physical activity, smoking, alcohol and drug use) and nutritional habits were questioned with the questionnaire form.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Icer MA, Yildiran H, Sahinarslan A, Topal S. Effects of Omega-3 Fatty Acid Supplementation on Serum Fetuin-A Levels in Patients With Coronary Artery Disease. Food Sci Nutr. 2025 Jun 18;13(6):e70460. doi: 10.1002/fsn3.70460. eCollection 2025 Jun. PMID 40538988